CLINICAL TRIAL: NCT05152316
Title: Inflammatory Markers and Surfactant Proteins in Preterm Infants at Risk of Developing Chronic Lung Disease: an Observational Study
Brief Title: The Baby Lung Study
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 138731
Record Dates: First submitted 2021-11-05; First posted 2021-12-09 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Bronchopulmonary Dysplasia; Neonatal Disease
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Infant, Newborn, Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — This is an observational study and no additional interventions will be done except for those that are standard care. Blood and tracheal aspirates will be taken to assess the surfactant protein levels and inflammatory markers including cell counts and cytokine levels.

SUMMARY:
The introduction of exogenous surfactant therapy has significantly improved the mortality in preterm infants born between 23- and 28-weeks of gestation. However, the therapy has not affected the prevalence of sequelae such as bronchopulmonary dysplasia [BPD] and it may be argued that it has actually increased. BPD is a lung condition that affects up to 40% of premature babies born between 23 and 28 weeks gestational age. The prevalence of BPD decreases with increasing gestational age but can affect infants born at term who have required mechanical ventilation. It is most commonly defined based on the need for oxygen past 36 weeks post-menstrual age [PMA]. The pathogenesis of BPD is multifactorial and involves a complex balance between the underdeveloped lungs, infection, inflammation, oxygen toxicity and ventilator induced injury.

In this study the investigators aim to develop a greater understanding of the interactions between the inflammatory markers present in endotracheal aspirates [ETA] and serum of preterm infants and surfactant components (including surfactant protein D-SP-D levels) in the lungs and in the serum of preterm ventilated infants.

The investigators aim to recruit infants born between 23+0 and 29+6 weeks of gestation at University College London Hospital admitted to the neonatal unit, who are at risk of developing respiratory distress syndrome [RDS] and progression to BPD. The investigators plan to study the correlation between the concentrations of surfactant components (in particular SP-D) and inflammatory markers in infants across the range of gestations specified. In order to do this, the investigators will obtain gastric aspirates, endotracheal aspirates [ETA] and blood samples at birth, 24hrs and days 2 through to day 7 from participants. ETA will only be obtained if the infants are intubated and ventilated, collected by a standard technique routinely used in nursing care of ventilated babies using 1-2mls of saline.ETA and blood samples will then be analysed for levels of surfactant proteins in particular SP-D and inflammatory and immunological markers [cell counts of neutrophils, macrophages, MMPs, neutrophil elastase, IL-8, IL-6, IL 11 and IL-1]. This will allow us to map the influence of SP-D on pro and anti-inflammatory markers that have a role in the inflammatory component of BPD in these infants.

Clinical data will also be collected at specified time points correlating with the plasma, gastric aspirates and endotracheal aspirates. The investigators aim to correlate clinical ventilatory parameters, infection factors and maternal factors with the inflammatory and surfactant protein profiles. In addition, the investigators will apply the international neonatal consortium Neonatal Adverse severity scores to gain a better understanding of the baseline incidence of adverse events in premature infants that are admitted to a neonatal unit.

ELIGIBILITY:
Inclusion Criteria:

. Preterm infants born between 23 weeks and 0 days and 30 weeks and 0 days gestation.

Exclusion Criteria:

* Congenital anomalies i.e any major antenatal diagnosed congenital abnormalities such as congenital heart disease, suspected or known chromosomal abnormalities.
* Infants not born at UCLH where baseline data and samples cannot be collected

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born between 23 + 0 weeks post menstrual age and 30 weeks post menstrual age.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
To analyses the profile of surfactant protein D in preterm infants at risk of bronchopulmonary dysplasia. | 24 months
  To measure the surfactant protein D levels in gastric and tracheal aspirates and plasma samples taken at birth, 24hrs, 48hrs, 72hrs, 96hrs, D7 of life and 36weeks post menstrual age if still intubated.
Characterise the inflammatory cell profile in preterm infant at high risk of developing bronchopulmonary dysplasia. | 24 months
  To analyse the gastric and tracheal aspirates and plasma samples taken at birth, 24hrs, 48hrs, 72hrs, 96hrs, D7 of life and 36weeks post menstrual age if still intubated for cell counts (macrophages and neutrophils) to better understand the correlation with SP-D over a period of time.
Characterise the cytokine profile in preterm infants at high risk of developing bronchopulmonary dysplasia. | 24 months
  To analyse the gastric and tracheal aspirates and plasma samples taken at birth, 24hrs, 48hrs, 72hrs, 96hrs, D7 of life and 36weeks post menstrual age if still intubated for pro- and anti-inflammatory cytokines to better understand the correlation with SP-D over a period of time.
To understand the incidence of adverse events in preterm infants at risk of developing bronchopulmonary dysplasia. | 24 months
  To apply the Neonatal Adverse Events Severity Score developed by the International Neonatal Consortium to better evaluate the incidence of adverse events in this vulnerable population.

SECONDARY OUTCOMES:
Association of inflammatory profile and surfactant components with clinical parameters. | 24 months
  To study the association of the inflammatory profile and concentration of surfactant components with clinical factors comprising of baseline factors, such as infant sex, ethnicity, administration of antenatal steroids, evidence of maternal sepsis/chorioamnionitis, and treatment factors, such as ventilator settings and tracheal colonisation.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Clark, Professor, Study Chair — University College, London; Reena Bhatt, Dr, Principal Investigator — University College, London
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data gathered will be the property of University College London and will not be shared with other research groups.